CLINICAL TRIAL: NCT06297499
Title: Timing of Ondansetron Use for Maximum Efficacy in Preventing Pruritus in Patients Undergoing Cesarean Section Under Spinal Anesthesia with Preservative Free Morphine.
Brief Title: Ondansetron Use for Preventing Pruritus in Patients Undergoing Cesarean Section
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Justin Hruska, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-22-07-4803
Record Dates: First submitted 2024-02-13; First posted 2024-03-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pruritus Caused by Drug
Keywords: Cesarean Section; Intrathecal Morphine; Ondansetron
MeSH Terms: interventions — Ondansetron; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient will be unaware of their grouping allotment. The outcomes assessor will be unaware of the patient grouping allotment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group 1. Pre-Intrathecal (Experimental): Patients will receive an IV solution of 8mg ondansetron (4ml) within 30 minutes of the standard-of-care anesthetic treatment (intrathecal morphine administration) followed by a placebo treatment of an IV solution of 4ml 0.9% saline administered at the time of umbilical cord clamping.
  Interventions: Drug: Ondansetron 8mg
- Treatment Group 2 Cord clamping (Active Comparator): Patients will receive a placebo treatment of an IV solution of 4ml 0.9% saline administered within 30 minutes of the standard-of-care anesthetic treatment (intrathecal morphine administration) followed by an IV solution of 8mg ondansetron (4ml) administered at the time of umbilical cord clamping.
  Interventions: Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Ondansetron 8mg — administration of an IV solution of 8mg ondansetron (4ml)
  Other Names: Placebo- 4ml of 0.9% IV saline

SUMMARY:
Opioids are often added with a local anesthetic to enhance the duration and quality of spinal anesthesia for cesarean delivery patients. However, spinal opioids are associated with a wide variety of side effects such as nausea, vomiting, (N/V) and pruritus (itching). The occurrence of pruritus can vary between 30% and 100% making pruritus the most common side-effect of intrathecal opioids and this rate is even higher in pregnant patients. Pruritus may require treatment which can be ineffective or sometimes reverse the analgesic effect of the opioids. Ondansetron is a safe and very commonly used Serotonin receptor antagonist treatment for local anesthetic opioid-induced pruritus used in pregnancy. The effect of different administration times of ondansetron in reducing pruritus or N/V in cesarean section (CS) cases has not been extensively studied and thus, this prospective study can help guide future clinical management of side effects caused by spinal intrathecal morphine administration.

DETAILED DESCRIPTION:
Opioids are often added with a local anesthetic to enhance the duration and quality of spinal anesthesia for cesarean delivery patients. However, spinal opioids are associated with a wide variety of side effects such as nausea, vomiting, (N/V) and pruritus (itching). The occurrence of pruritus can vary between 30% and 100% making pruritus the most common side-effect of intrathecal opioids and this rate is even higher in pregnant patients. Pruritus may require treatment which can be ineffective or sometimes reverse the analgesic effect of the opioids. Ondansetron is a safe and very commonly used Serotonin receptor antagonist treatment for local anesthetic opioid-induced pruritus used in pregnancy. The effect of different administration times of ondansetron in reducing pruritus or N/V in cesarean section (CS) cases has not been extensively studied and thus, this prospective study can help guide future clinical management of side effects caused by spinal intrathecal morphine administration.

The primary aim of this study is to observe in a randomized double-blinded trial if the timing of prophylactic administration of intravenous ondansetron can reduce the incidence and severity of intrathecal morphine-induced pruritus in patients undergoing Cesarean section (CS). The secondary aim is to establish the effect of intravenous ondansetron given at different time intervals following CS for postoperative nausea and vomiting (PONV). The primary study hypothesis is that patients receiving prophylactic intravenous ondansetron (15-30 minutes prior to intrathecal morphine) will experience a lower incidence and severity of intrathecal morphine-induced pruritus than patients receiving ondansetron administered at the time of umbilical cord clamping. The secondary study hypothesis is that CS patients receiving intravenous ondansetron 15-30 minutes prior to intrathecal morphine will have less nausea and vomiting than patients receiving ondansetron administered at the time of umbilical cord clamping.

As the effect of prophylactic administration of ondansetron in reducing pruritus or Nausea/Vomiting in cesarean section (CS) cases has not been studied and thus, this prospective study may help guide future clinical management of side effects caused by intrathecal morphine administration.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1-3
2. Adult parturient (18 -50 years of age) scheduled to undergo elective cesarean delivery under spinal anesthesia
3. Patients must be willing and cognitively able to give written informed study consent

Exclusion Criteria:

1. Patients with an ASA physiological assessment greater than grade 3
2. Allergies to local anesthetics, opioids, or ondansetron
3. Coagulopathies precluding provision of spinal anesthesia
4. Pre-eclampsia with severe features
5. Eclampsia
6. Pre-intrathecal pruritus
7. Psychiatric or language deficiencies affecting assessment of pain
8. Insufficient understanding of the pain scoring system
9. Patients who receive any other regional anesthesia techniques
10. Patients on higher than a 100mg of daily morphine equivalent
11. Cardiac issues that would preclude spinal anesthesia (Congestive heart failure, Mitral or Aortic valve pathology.
12. Confounding neural issues that would preclude spinal anesthesia.
13. Coadministration of drugs that would potentially interact with ondansetron. Including Apomorphine, Phenytoin, Carbamazepine, Rifampicin, Tramadol and Chemotherapy drugs.
14. Coadministration of drugs that would potentially prolong QTc interval. Including Antiarrhythmic, Antidepressants, Antipsychotics, and the following list of medications.

    a. Levofloxacin, Ciprofloxacin, Gatifloxacin, Moxifloxacin, Clarithromycin, Erythromycin, Ketoconazole, Itraconazole, Cisapride, Sumatriptan, Zolmitriptan, Arsenic, Dolasetron, Methadone
15. Coadministration of drugs that would potentially lead to the development of serotonin syndrome. Including the following:

    a. Selective serotonin reuptake inhibitors, Serotonin and norepinephrine reuptake inhibitors, antidepressants, carbamazepine , valproic acid, triptans, Chronic pain medications prior to procedure (Fentanyl, Hydrocodone, Meperidine, Oxycodone, tramadol),Lithium, dextromethorphan, Linezolid and Ritonavir
16. Patients having the following

    1. Patients known to have hypersensitivity (e.g., anaphylaxis) to ondansetron or any components of the formulation
    2. Concomitant use of apomorphine
    3. History of QTc interval prolongation (QTc >440) and Torsade de Pointes
    4. Serotonin syndrome
    5. Phenylketonuric patients
    6. Concurrent use of selective serotonin reuptake inhibitors (SSRIs) and serotonin and noradrenaline reuptake inhibitors (SNRIs)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pruritus parameters in Post anesthesia Care Unit (PACU) | Assessment during 1st post-operative hour in PACU
  Patient Assessment (patient questionnaire): Pruritus occurrence (Yes or no) and anatomical location of Pruritus of occurrence, Severity of Pruritus- Likert scale choices from (Not present, Mild, Moderate, Severe, Unbearable) severity
Pruritus severity in Post anesthesia Care Unit (PACU) | Assessment during 1st post-operative hour in PACU
  Severity of Pruritus- Likert scale choices from (Not present, Mild, Moderate, Severe, Unbearable) severity
Pruritus parameters PACU | Assessment during 24 hours post-operative period
  Patient Assessment (patient questionnaire): Pruritus occurrence (Yes or no) and anatomical location of pruritus location
Pruritus severity PACU | Assessment during 24 hours post-operative period
  Patient Assessment (patient questionnaire): Pruritus Severity: Likert scale: choice of (Not present, Mild, Moderate, Severe, Unbearable)
Rescue Pruritus Treatment medication | Measured in the 24 hour period from initial study treatment (30 minute period before intrathecal morphine administration.
  Patient Assessment questionnaire: If rescue Pruritus treatment was required (YES/NO) and if so specific medication type and dose amount of medication
Nausea PACU | Assessment every 15 minutes for 1 hour
  Patient Assessment questionnaire: Severity of Nausea- Likert scale: choice of (Not present, Mild, Moderate, Severe, Unbearable)
Nausea Post PACU | our period after patients left PACU from initial study treatment (30 minute period before intrathecal morphine administration.
  Patient Assessment questionnaire: Severity of Nausea- Likert scale: choice of (Not present, Mild, Moderate, Severe, Unbearable)

SECONDARY OUTCOMES:
Post-operative Pain | Taken while patient in PACU at 0 minutes, 15 minutes, 30 minutes, 45 minutes and 60 min. Post PACU patient assessment at at 8 hours, 16 hours, 24 hours post-operative period
  Patient assessment questionnaire: Visual analog pain scale (VAS) measuring scores from 0 (no pain)-10 (worst pain) at rest

OTHER OUTCOMES:
Peripheral oxygen saturation- Mother | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient Peripheral blood oxygen saturation (percentage %) via a pulse oximeter
Peripheral oxygen saturation- Infant | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient Peripheral blood oxygen saturation (percentage %) via a pulse oximeter
Heart rate- Mother | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient heart rate (beats per minute) via a pulse oximeter
Heart rate- Infant | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient heart rate (beats per minute) via a pulse oximeter
Blood pressure Mother | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient blood pressure (Diastolic/Systolic pressure mm/Hg) 0
Blood pressure- Infant | At Delivery, then at 30 minutes, 60 minutes, 90 minutes, 2 hours, 8 hours,16 hours, 24 hours post-delivery
  Clinical Measurement of patient blood pressure (Diastolic/Systolic pressure mm/Hg) 0
Electrocardiogram (ECG ) Mother | Within 2 hours of birth.
  ECG parameters (ECG QT intervals) interpreted by a by a trained Cardiologist
ECG Infant | Within 2 hours of birth.
  ECG parameters (ECG QT intervals) interpreted by a by a trained Cardiologist

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Medical Center- Hutzel Women's Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No